CLINICAL TRIAL: NCT07075549
Title: Cross-cultural Validation of the French Version of the Lymphedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphedema (Lymph-ICF-LL) and Responsiveness of the Dutch Version of the Lymph-ICF-LL
Brief Title: Psychometric Properties of a Lymphedema-specific Quality of Life Questionnaire in Lower Limb Lymphedema
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: CHU UCL Namur (Unknown)
Responsible Party: Sponsor
Other Study IDs: S67308
Record Dates: First submitted 2025-07-08; First posted 2025-07-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Lymphedema Lower Extremity
Keywords: Reliability; Validity; Responsiveness; Quality of Life; Questionnaire; Lymphedema; Lower Limb
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Native French speaking patients with stable lower limb lymphedema in the maintenance phase: Native French speaking patients with stable lower limb lymphedema in the maintenance phase were included for the reliability, validity and responsiveness of the French Lymph-ICF-LL
  Interventions: Other: Maintenance phase of Decongestive Lymphatic Therapy
- Native French speaking patients with lower limb lymphedema which are treated in the intensive phase: Native French speaking patients with lower limb lymphedema who received treatment in the intensive phase were included for the responsiveness of the French Lymph-ICF-LL
  Interventions: Other: Intensive phase of Decongestive Lymphatic Therapy
- Native Dutch speaking patients with stable lower limb lymphedema in the maintenance phase: Native Dutch speaking patients with stable lower limb lymphedema in the maintenance phase were included for the responsiveness of the Dutch Lymph-ICF-LL
  Interventions: Other: Maintenance phase of Decongestive Lymphatic Therapy
- Native Dutch speaking patients with lower limb lymphedema which are treated in the intensive phase: Native Dutch speaking patients with lower limb lymphedema who received treatment in the intensive phase were included for the responsiveness of the Dutch Lymph-ICF-LL
  Interventions: Other: Intensive phase of Decongestive Lymphatic Therapy

INTERVENTIONS:
Other: Maintenance phase of Decongestive Lymphatic Therapy — Patients with lower limb lymphedema in the maintenance phase of decongestive lymphatic therapy (with compression garments) were included
  Groups: Native Dutch speaking patients with stable lower limb lymphedema in the maintenance phase; Native French speaking patients with stable lower limb lymphedema in the maintenance phase
Other: Intensive phase of Decongestive Lymphatic Therapy — Patients with lower limb lymphedema who are treated in the intensive phase of Decongestive Lymphatic Therapy (with multilayer bandages) were included
  Groups: Native Dutch speaking patients with lower limb lymphedema which are treated in the intensive phase; Native French speaking patients with lower limb lymphedema which are treated in the intensive phase

SUMMARY:
The goal of this observational study is to cross-validate the Lymphedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphedema (Lymph-ICF-LL) in French and to investigate the responsiveness of the original Dutch Lymph-ICF-LL questionnaire in patients with lower limb lymphedema. The main questions it aims to answer are:

1. The reliability of the French Lymph-ICF-LL
2. The validity of the French Lymph-ICF-LL
3. The responsiveness of the original Dutch Lymph-ICF-LL

Participants are asked to complete questionnaires (Lymph-ICF-LL, Short Form-36, Global Perceived Effect Scale, questionnaire about the face and content validity) at two time points.

DETAILED DESCRIPTION:
1. For reliability of the French Lymph-ICF-LL questionnaire:

   Native French speaking patients with stable lower limb lymphedema (LLL) (= in the maintenance phase of the treatment and no intensive multicomponent bandaging is required) are asked to complete the Lymph-ICF-LL questionnaire twice with an interval of 1-2 days in between.

   For the test-retest reliability following outcomes are calculated: Intraclass Correlation Coefficient(2,1), standard error of measurement and the smallest real difference.

   For internal consistency the Cronbach's alpha is calculated for the first completion of the questionnaire.
2. For the validity of the French Lymph-ICF-LL questionnaire, the construct validity, face and content validity are determined.

   2.1: For construct validity (=convergent and divergent validity), patients with stable lower limb lymphedema are asked to additionally complete the 36-item Short-Form Health survey (=health-related quality of life questionnaire) together with the first completion of the Lymph-ICF-LL questionnaire. For convergent validity, hypotheses are formulated about significant correlations between domains of the 36-item Short-Form Health survey (=SF-36) and domains of the Lymph-ICF-LL questionnaire which are expected to evaluate a similar construct: 'Physical functioning' of SF-36 and 'general tasks/household', 'mobility', 'life domains/social life' of the Lymph-ICF-LL; 'Role limitations due to physical health problems' of SF-36 and 'General tasks/household' of Lymph-ICF-LL; 'Bodily pain' of SF-36 and 'Physical function' of Lymph-ICF-LL; 'Social functioning' of SF-36 and 'Life domains/ social life' of Lymph-ICF-LL; 'Role limitations due to personal or emotional problems' of SF-36 and 'Mental function' of Lymph-ICF-LL; 'Mental health' of SF-36 and 'Mental function' of Lymph-ICF-LL. For divergent validity, hypotheses are formulated about weak or non-significant correlations between domains of the SF-36 and Lymph-ICF-LL: 'Physical functioning' of SF-36 and 'Mental function' of Lymph-ICF-LL; 'Role limitations due to personal or emotional problems' of SF-36 and 'Physical function' Lymph-ICF-LL; 'Mental health' of SF-36 and 'General tasks/household', 'Mobility', 'Life domains/social life' of Lymph-ICF-LL. These hypotheses were also used in previous published research of the validation of the original Dutch Lymph-ICF-LL questionnaire. Spearman rank correlation coefficients were calculated for this purpose.A correlation coefficient below .25 represent no to a little relationship, a value between .25 and .50 indicates a low to fair relationship, a value between .50 and .75 is interpreted as a moderate to good relationship and a value above or equal to .75 as a strong relationship.

   2.2 For face and content validity, patients with stable LLL are asked to complete an additional questionnaire about clarity and completeness of the Lymph-ICF-LL questionnaire: "Was each question of the Lymph-ICF-LL understandable? (yes/no)", "Was the scoring system clear? (yes/no)", "Were all complaints related to your lymphedema mentioned in the questionnaire? (yes/no)" and "Where there any questions of which you thought they were not relevant for lymphedema? (yes/no)". If patients answered 'no', they could clarify their answer in an open field.
3. For the responsiveness of the French and Dutch Lymph-ICF-LL, internal and external responsiveness is evaluated in patients with stable LLL and in patients who are treated in the intensive phase with multicomponent bandages. For internal responsiveness, patients with stable LLL have to complete the Lymph-ICF-LL questionnaire twice with an interval of 2 months. Patients treated in the intensive phase have to complete the questionnaire at the start of the intensive phase and 1 month after the end of the intensive phase. The Wilcoxon signed rank test is determined to evaluate if there is a significant difference between the total and subdomain scores of two completions in patients in the intensive phase and not in patients with LLL. For the external responsiveness, all patients are asked to complete the Global Perceived effect scale (GPE) together with the second completion of the Lymph-ICF-LL questionnaire. In this GPE questionnaire patient are asked to rate their perceived change in lymphedema-specific quality of life in general and concerning the subdomains of the Lymph-ICF-LL on a 7-point Likert-scale: 1=completely recovered, 2=much better, 3= a little better, 4= unchanged, 5= a little worse, 6= much worse, 7= worse than ever. Patients who give score 1 and 2 are labeled as responders, with score 3-5 as non-responders and with scere 6-7 as negative responders. The Wilcoxon signed rank test was determined between the total and subdomain scores in the positive, negative and non responder groups. Additionally spearman rank correlations coefficients are calculated between the change in total and subdomain scores and the GPE-score. The minimal clinically important difference are calculated with the anchor-based method: descriptive statistics of the change in total and subdomain scores of the Lymph-ICF-LL are determined in patients who indicated on the GPE that the lymphedema-specific quality of life was much improved or much worsened.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary lymphedema at the lower limb(s), i.e. a difference of ≥5% in volume between the two sides or a lymphoscintigraphy which shows at least 2 minor criteria or 1 major criterion or presence of indocyanine green (ICG) dermal backflow
* Unilateral/bilateral lymphedema
* Lymphedema stage 1, 2a, 2b or 3
* Lymphedema is present >3 months
* Chemotherapy and radiotherapy was finished >3 months ago
* Native French-speaking or Dutch-speaking for study about the French or Dutch Lymph-ICF-LL, respectively
* During the study patients are in the maintenance phase and not in the intensive phase (for the reliability/validity/responsiveness); patients receive intensive treatment in the hospital (for the responsiveness)
* Given informed consent to participate
* >18 years old

Exclusion Criteria:

* Not able to read or fully understand the French or Dutch language for study about the French or Dutch Lymph-ICF-LL, respectively
* For the reliability and validity and for part of the responsiveness: first treatment for lymphedema < 6 months ago and an intensive phase is planned or needed according to a specialized caregiver in treating lymphedema
* <18 years old
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower limb lymphedema are treated with decongestive lymphatic therapy and are either in the intensive phase or in the maintenance phase. Patients in both phases are included in this study.
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Reliability of the French Lymph-ICF-LL questionnaire (test-retest) | Baseline and 1-2 days later
  Following aspects were assessed to investigate the reliability of the French Lymph-ICF-LL:
  Test-retest relative reliability Patients completed the Lymph-ICF-LL two times with an interval of 1-2 days. The total score and subdomain scores are calculated: (sum of scores divided by the number of completed questions)*10. This results in a score between 0 and 100 in which 0 reflects a better lymphedema-specific quality of life and 100 a worse lymphedema-specific quality of life. The intraclass correlation coefficient (2,1) (ICC) is calculated between the first and second completion. An ICC above .90 is interpreted as excellent relative reliability, an ICC between .75 and .90 as good, an ICC between .50 and .75 as moderate and an ICC below .50 as poor relative reliability.
Reliability of the French Lymph-ICF-LL questionnaire (standard error of measurement) | Baseline and 1-2 days later
  Standard error of measurement (SEM) reflects absolute reliability between the total and subdomain scores of the Lymph-ICF-LL questionnaires at baseline and 1-2 days later. The SEM is calculated with the square root of mean square error determined by ANOVA.
Reliability of the French Lymph-ICF-LL questionnaire (smallest real difference) | Baseline and 1-2 days later
  Smallest Real Difference (SRD) between the total and subdomain scores of the two Lymph-ICF-LL questionnaire completions at baseline and 1-2 days later was calculated by 1.96 multiplied by SEM and square root of 2.
Reliability of the French Lymph-ICF-LL questionnaire | Baseline (first completion of the Lymph-ICF-LL questionnaire)
  Internal consistency with Cronbach's alpha of the different domains and total score. A Cronbach's alpha between .70 and .90 is considered as a good internal consistency

SECONDARY OUTCOMES:
Face and content/floor & ceiling effects of the French Lymph-ICF-LL | Baseline
  A self-developed questionnaire was completed by the patients with stable lower limb lymphedema with questions about the clarity of the scoring system and questions, the completeness and redundancy of the questions of the Lymph-ICF-LL. Frequency of the minimum and maximum score was reported to evaluate floor (frequency of score 0 on the total score and subdomain scores of the Lymph-ICF-LL questionnaire) and ceiling (frequency of score 100 on the total score and subdomain scores of the Lymph-ICF-LL questionnaire) effects, respectively.
Construct validity of the Lymph-ICF-LL | Baseline
  Hypothesis about which domains of the lymph-ICF-LL would be highly correlated with certain domains of the short form health survey with 36 items (SF-36) were formulated to assess convergent validity. To evaluate discriminant validity hypothesis were formulated on which domains of the lymph-ICF-LL would have a weak correlation with certain domains of the SF-36. The SF-36 was completed together with the first completion of the Lymph-ICF-LL by patients with stable lower limb lymphedema. For both the SF-36 and Lymph-ICF-LL questionnaires scores varied between 0 and 100. However, for the SF-36 a scores closer to zero reflect a worse quality of life, while for the Lymph-ICF-LL scores closer to zero reflect a better lymphedema-specific quality life.
Internal responsiveness of the Lymph-ICF-LL | At start of the intensive phase and 1 month after the end of the intensive phase (patients receiving intensive treatment) or at baseline and 2 months later (patients with stable lower limb lymphedema)
  Internal responsiveness evaluates the ability of the questionnaire to have different results over a particular timeframe. For this purpose two groups of patients were included: one group where a change in lymphedema-specific quality of life can be expected (patients receiving intensive treatment) and one group where no change in lymphedema-specific quality of life is expected (patients with stable lower limb lymphedema). The Lymph-ICF-LL had to be completed at two time points (see Time Frame). A score closer to zero reflects a better lymphedema-specific quality of life and a score closer 100 reflects a worse lymphedema-specific quality of life.
External responsiveness | Start of the intensive phase and 1 month after the end of the intensive phase (patients receiving intensive treatment) or baseline an 2 months later (patients with stable lower limb lymphedema in the stable phase)
  = extent to which the change on the Lymph-ICF-LL is related to the change on a reference measure of a person's health status over a certain time period. 2 groups of patients are included: 1 group in which a change in lymphedema-specific quality of life is expected (patients receiving intensive treatment) and 1 group in which no change in lymphedema-specific quality of life is expected (patient with stable lower limb lymphedema). The Lymph-ICF-LL is completed at 2 time points (see Time Frame). Additionally, the global perceived effect scale (GPE) was completed at the second time point in which patients have to evaluate on a 7-point Likert scale their current health status in comparison with an earlier defined timepoint. 1=completely recovered, 2=much better, 3=a little better, 4=unchanged, 5=a little worse, 6=much worse, 7=worse than ever. Patients were divided in groups. Scores 1,2= positive responder, scores 3,4,5= non-responder, scores 6,7= negative responder

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - UZ Leuven and KU Leuven, Leuven
  - CHU UCL Namur site Godinne, Yvoir
- Hôpital Cognacq-Jay, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available on reasonable request.